CLINICAL TRIAL: NCT00376363
Title: Ahmed Versus Baerveldt Comparison Study
Acronym: ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Eye Institute (NEI) (NIH); Research to Prevent Blindness (Other)
Responsible Party: Principal Investigator, Donald L. Budenz, Study Chairman, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20057138; P30EY014801 (NIH)
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Glaucoma
Keywords: glaucoma; Ahmed implant; Baerveldt implant
MeSH Terms: conditions — Glaucoma | interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ahmed implant,1 (Active Comparator): Ahmed glaucoma drainage implant for intraocular pressure control
  Interventions: Device: Ahmed implant
- Baerveldt implant (Active Comparator): Baerveldt glaucoma drainage implant for intraocular pressure control
  Interventions: Device: Baerveldt implant

INTERVENTIONS:
Device: Ahmed implant — placement of glaucoma drainage device to control intraocular pressure
  Other Names: Ahmed fp7
  Arms: Ahmed implant,1
Device: Baerveldt implant — placement of glaucoma drainage device to control intraocular press
  Other Names: Baerveldt 350
  Arms: Baerveldt implant

SUMMARY:
The objective of this study is to compare the long-term safety and efficacy of the Ahmed and the Baerveldt implants in patients who are undergoing aqueous shunt implant surgery for glaucoma. One eye of eligible patients will be randomized. Outcome measures include intraocular pressure, visual acuity, visual field, number of glaucoma medications, glaucoma reoperations, and complications, including suprachoroidal hemorrhage, endophthalmitis, choroidal effusion, diplopia, corneal edema, and shunt/tube erosion.

DETAILED DESCRIPTION:
Background and Significance

Aqueous shunt devices have traditionally been reserved for treatment of only the most refractory glaucomas. However, more recent studies have reported favorable results in comparison with trabeculectomy in medically uncontrolled glaucomas at lower risk of filtration failure. Consequently, aqueous shunt devices have been used increasingly in glaucoma drainage surgery.

There are two principal designs of implant in common use, the Ahmed glaucoma valve implant (New World Medical, Los Ranchos, CA, USA and the Baerveldt implant (Advanced Medical Optics, Santa Ana, CA, USA).

Having both evolved from the Molteno, the Ahmed and Baerveldt devices have in common a tube portion that drains aqueous humor from the anterior chamber to a plate that is implanted on the equatorial sclera. The size of plate determines the surface area of the drainage bleb.

The Ahmed and Baerveldt implants differ in two major respects. Firstly, the plate surface area of the Baerveldt 350 implant is almost double that of the Ahmed (185 mm2). Secondly, the Ahmed has a flow-restrictor that limits early hypotony without the need for additional external ligation.

We propose a randomized prospective clinical trial comparing the long-term safety and efficacy of the Ahmed glaucoma valve implant (FP-7) with the 350-mm2 Baerveldt implant (101-350) for surgical control of secondary glaucoma and primary glaucoma in eyes that have undergone previous ocular surgery.

Objective

The objective of this study is to compare the long-term safety and efficacy of the Ahmed FP-7 implant and the 350-mm2 Baerveldt implant in patients who are undergoing aqueous shunt implant surgery. Patients who qualify for the study are randomized to receive either an Ahmed FP-7 or Baerveldt BG-101-350 implant. Only one eye of a patient may be enrolled in the study.

Outcome discrimination between the two treatment groups will be made using typical measures of visual function (visual acuity and visual field), intraocular pressure, number of glaucoma medications, and glaucoma reoperations. Emphasis will also be placed on complication rates, including suprachoroidal hemorrhage, endophthalmitis, choroidal effusion, diplopia, corneal edema, and shunt/tube erosion.

Assignment

Since the purpose of this study is to compare the safety and efficacy of two surgical procedures used in the management of glaucoma, randomization techniques are used to assure an unbiased treatment assignment to patients.

Stratification:

Patients will be stratified by clinical center. At each Clinical Center, half of the patients will receive an Ahmed and half will receive a Baerveldt implant. Randomization takes place at the time the patient is enrolled in the study after informed consent is obtained.

Randomization:

A permuted variable block randomization scheme stratified by clinical center and type of glaucoma will be performed.

The following scenarios will constitute a failure in the ABC Study for the purposes of survival analysis:

* IOP > 21mmHG or < 6mmHg on 2 consecutive study visits at visits > 3 months
* IOP reduced by < 20% on 2 consecutive study visits at visits > 3 months
* Reoperation for glaucoma
* Loss of light perception vision
* Removal of implant for any reason

Clinical Procedures

Visual Acuity

Visual acuity is an important outcome variable in the ABC Study. Visual acuity is measured before pupil dilation, tonometry, gonioscopy, or any other technique that could affect vision. Refraction is performed prior to formal measurement of visual acuity by either technique at the Qualifying Assessment and at the annual follow-up visits. Snellen visual acuity is measured at the Qualifying Assessment and at every follow-up visit.

Subjective refraction must be performed at the Qualifying Assessment and at the annual follow-up visits in order to determine best-corrected visual acuity. It is permissible to use a phoropter or trial frame to determine best-corrected Snellen visual acuity.

Slit Lamp Biomicroscopy Conjunctiva examination Cornea examination An assessment is made of the position and length of the tube in the eye. Anterior Chamber examination Iris examination Lens examination Tonometry Goldmann applanation tonometry is used to measure the intraocular pressure, except when irregular corneal astigmatism, corneal scarring, or corneal edema precludes accurate readings. In these cases, the Tono-Pen (Mentor) is used. The intraocular pressure is measured prior to pupillary dilation. Whenever possible, the intraocular pressure should be checked at the same time of the day as the Qualifying Assessment to minimize the effect of diurnal fluctuation The Tono-Pen (Mentor) is used in cases of corneal edema, corneal scarring, or irregular corneal astigmatism.

Central corneal thickness will be measured in each eye, by ultrasound pachymetry. A minimum of 5 measurements will be taken and the lowest recorded.

Motility Evaluation Gonioscopy Ophthalmoscopy Perimetry Visual field assessment is an important outcome measure in the ABC Study. Quantitative automated perimetry is performed using the Humphrey Field Analyzer. Visual field testing is performed before tonometry, gonioscopy, or any other technique that could affect vision. A visual field should be attempted in any eye that has sufficient vision to permit finger counting at two feet. Eyes with poor central vision may have an intact, off-center island of vision which may be measured with perimetry.

For the ABC Study, a 24-2 threshold test is performed in all patients using a size III white stimulus. Visual field testing may be performed with the Swedish Interactive Thresholding Algorithm (SITA) or full threshold strategy, but the same testing strategy must be used throughout the duration of the study. The pupil diameter should be 3 mm or greater before visual field testing is undertaken, and this may require pharmacologic dilation. Standardized refraction is performed to determine the patient's distance refraction and best-corrected visual acuity prior to visual field testing. The age appropriate plus lens is added to the distance refraction. Patient education is provided, and the instrument is set up for the test. The technician should monitor the patient during testing. Visual fields are performed preoperatively (within one month of enrollment in the study) and annually thereafter. Copies of all visual fields are faxed to the Statistical Coordinating Center for evaluation.

Surgical Procedures

The type of anesthesia is at the surgeon's discretion.

Conjunctival Flap:

An Ahmed FP-7 is used in all cases and implantation is performed in the superotemporal quadrant. A limbus-based or fornix-based conjunctival flap may be used depending on the surgeon's preference. Sufficient exposure is obtained in the superotemporal quadrant to permit placement of the Ahmed plate. A corneal traction suture or episcleral traction suture may be used to rotate the globe inferonasally to improve exposure.

Priming the Implant

A 28- or 30- gauge cannula is used to prime the Ahmed valve. Occlusion of the tube with a ligature is not permitted.

Attachment of Episcleral Plate:

The Ahmed plate is sutured to the sclera at a measured distance of 8 - 10 mm posterior to the limbus using the two fixation holes on the plate. The type of nonabsorbable suture used is of the surgeon's choice.

Preparation of Tube:

The tube is trimmed bevel-up to extend 2 to 3 mm into the anterior chamber.

Insertion of Tube into the Anterior Chamber:

A 23-gauge needle is used to enter the anterior chamber at the posterior limbus parallel to the iris plane. The Ahmed tube is inserted through this entry incision and should be well positioned in the anterior chamber away from the corneal endothelium and just above the iris. A 23-gauge needle produces an adequate entry incision for the tube without causing aqueous leakage around the tube.

Coverage of Tube:

A donor patch graft composed of donor sclera, donor cornea, or pericardium is used to cover the limbal portion of the tube. The suture selected to fixate the patch graft is of the surgeon's choice.

Conjunctival Closure:

Tenon's and conjunctiva are reapproximated to the limbus. The suture used for the conjunctival closure is determined by the surgeon in keeping with his or her usual practice.

At the surgeons discretion, a viscoelastic of his or her choice may be inserted into the anterior chamber, especially if the anterior chamber shallows after balanced salt solution is inserted.

The use of intraoperative medications is at the surgeon's discretionBaerveldt Implantation The type of anesthesia is at the surgeon's discretion.

Conjunctival Flap:

A 350-mm2 Baerveldt is used in all cases and implantation is performed in the superotemporal quadrant. A limbus-based or fornix-based conjunctival flap may be used depending on the surgeon's preference.

Scleral Exposure:

Sufficient exposure is obtained in the superotemporal quadrant to permit placement of the Baerveldt plate. A corneal traction suture or episcleral traction suture may be used to rotate the globe inferonasally and improve exposure.

Insertion of Episcleral Plate:

The 350-mm2 Baerveldt plate may be positioned under or over the superior rectus and lateral rectus muscles, depending on the surgeon's usual practice. The implant is sutured to the sclera at a measured distance of 8 - 10 mm posterior to the limbus using the two fixation holes on the plate. The type of nonabsorbable suture used is of the surgeon's choice.

Occlusion of Tube:

The Baerveldt tube must be completely occluded in all cases in order to restrict aqueous flow to the plate until it becomes encapsulated. This is done to minimize the incidence of postoperative hypotony. The method of tube occlusion is left to the discretion of the surgeon. Ligation of the tube with a polyglactin suture near the tube-plate junction, ligation with a polypropylene suture which is inserted into the anterior chamber with the tube, or internal occlusion of the tube using a "rip-cord" technique have all been used effectively. A 30-gauge cannula is used to cannulate the end of the tube and confirm complete occlusion of the tube. Following tube occlusion, the surgeon may fenestrate the tube if desired. The method of tube fenestration is left to the discretion of the surgeon.

Preparation of Tube:

The tube is trimmed bevel-up to extend 2 to 3 mm into the anterior chamber.

Insertion of Tube into the Anterior Chamber:

A 23-gauge needle is used to enter the anterior chamber at the posterior limbus parallel to the iris plane. The Baerveldt tube is inserted through this entry incision and should be well positioned in the anterior chamber away from the corneal endothelium and just above the iris. A 23-gauge needle produces an adequate entry incision for the tube without causing aqueous leakage around the tube.

Coverage of Tube:

A donor patch graft composed of donor sclera, dura mater, or pericardium is used to cover the limbal portion of the tube. The suture selected to fixate the patch graft is of the surgeon's choice.

Conjunctival Closure:

Tenon's and conjunctiva are reapproximated to the limbus. The suture used for the conjunctival closure is determined by the surgeon in keeping with his or her usual practice.

The use of intraoperative medications is at the surgeon's discretion.

Multicenter clinical trials require an organizational structure that provides efficient operations and facilitates communication. The following resource centers work together in this study:

* Clinical Centers (CC)
* Statistical Coordinating Center (SCC)
* Safety and Data Monitoring Committee (SDMC)
* Steering Committee (SC)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years, inclusive.
* Glaucoma that is inadequately controlled on tolerated medical therapy with intraocular pressure greater than or equal to 18 mm Hg.
* Glaucoma drainage implant as planned surgical procedure.
* POAG with previous failed trabeculectomy or other intraocular surgery.
* Secondary glaucoma with or without previous intraocular surgery

Exclusion Criteria:

* Unwilling or unable to give consent or unwilling to accept randomization.
* Patient out of area and potentially unavailable for follow-up visits
* No light perception.
* Uveitis secondary to Juvenile Idiopathic Arthritis
* Previous cyclodestructive procedure or previous aqueous shunt device implanted in the same eye.
* Supero-temporal buckling or other external impediment to supero-temporal aqueous shunt implantation.
* Silicone oil-filled eyes or sufficient residual intraocular silicone oil to preclude supero-temporal aqueous shunt implantation.
* Vitreous sufficient to require a vitrectomy present in the anterior chamber at the time of surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2005-11; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Budenz, M.D.,M.P.H., Principal Investigator — University of North Carolina; Keith Barton, M.D., Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust; William J Feuer, M.S., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Bascom Palmer Eye Institute, Miami, Florida, United States

REFERENCES:
- [Background] Coleman AL, Hill R, Wilson MR, Choplin N, Kotas-Neumann R, Tam M, Bacharach J, Panek WC. Initial clinical experience with the Ahmed Glaucoma Valve implant. Am J Ophthalmol. 1995 Jul;120(1):23-31. doi: 10.1016/s0002-9394(14)73755-9. PMID 7611326
- [Background] Topouzis F, Coleman AL, Choplin N, Bethlem MM, Hill R, Yu F, Panek WC, Wilson MR. Follow-up of the original cohort with the Ahmed glaucoma valve implant. Am J Ophthalmol. 1999 Aug;128(2):198-204. doi: 10.1016/s0002-9394(99)00080-x. PMID 10458176
- [Background] Lloyd MA, Baerveldt G, Fellenbaum PS, Sidoti PA, Minckler DS, Martone JF, LaBree L, Heuer DK. Intermediate-term results of a randomized clinical trial of the 350- versus the 500-mm2 Baerveldt implant. Ophthalmology. 1994 Aug;101(8):1456-63; discussion 1463-4. doi: 10.1016/s0161-6420(94)31152-3. PMID 8058290
- [Background] Britt MT, LaBree LD, Lloyd MA, Minckler DS, Heuer DK, Baerveldt G, Varma R. Randomized clinical trial of the 350-mm2 versus the 500-mm2 Baerveldt implant: longer term results: is bigger better? Ophthalmology. 1999 Dec;106(12):2312-8. doi: 10.1016/S0161-6420(99)90532-8. PMID 10599663
- [Background] Wang JC, See JL, Chew PT. Experience with the use of Baerveldt and Ahmed glaucoma drainage implants in an Asian population. Ophthalmology. 2004 Jul;111(7):1383-8. doi: 10.1016/j.ophtha.2003.11.005. PMID 15234141
- [Background] Tsai JC, Johnson CC, Dietrich MS. The Ahmed shunt versus the Baerveldt shunt for refractory glaucoma: a single-surgeon comparison of outcome. Ophthalmology. 2003 Sep;110(9):1814-21. doi: 10.1016/S0161-6420(03)00574-8. PMID 13129882
- [Background] Nguyen QH, Budenz DL, Parrish RK 2nd. Complications of Baerveldt glaucoma drainage implants. Arch Ophthalmol. 1998 May;116(5):571-5. doi: 10.1001/archopht.116.5.571. PMID 9596491
- [Result] Barton K, Gedde SJ, Budenz DL, Feuer WJ, Schiffman J; Ahmed Baerveldt Comparison Study Group. The Ahmed Baerveldt Comparison Study methodology, baseline patient characteristics, and intraoperative complications. Ophthalmology. 2011 Mar;118(3):435-42. doi: 10.1016/j.ophtha.2010.07.015. Epub 2010 Oct 8. PMID 20932581
- [Result] Budenz DL, Barton K, Feuer WJ, Schiffman J, Costa VP, Godfrey DG, Buys YM; Ahmed Baerveldt Comparison Study Group. Treatment outcomes in the Ahmed Baerveldt Comparison Study after 1 year of follow-up. Ophthalmology. 2011 Mar;118(3):443-52. doi: 10.1016/j.ophtha.2010.07.016. Epub 2010 Oct 8. PMID 20932583
- [Result] Barton K, Feuer WJ, Budenz DL, Schiffman J, Costa VP, Godfrey DG, Buys YM; Ahmed Baerveldt Comparison Study Group. Three-year treatment outcomes in the Ahmed Baerveldt comparison study. Ophthalmology. 2014 Aug;121(8):1547-57.e1. doi: 10.1016/j.ophtha.2014.01.036. Epub 2014 Apr 24. PMID 24768240
- [Result] Budenz DL, Barton K, Gedde SJ, Feuer WJ, Schiffman J, Costa VP, Godfrey DG, Buys YM; Ahmed Baerveldt Comparison Study Group. Five-year treatment outcomes in the Ahmed Baerveldt comparison study. Ophthalmology. 2015 Feb;122(2):308-16. doi: 10.1016/j.ophtha.2014.08.043. Epub 2014 Oct 17. PMID 25439606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 276 patients were enrolled between November 2005 and April 2008: 143 in the Ahmed group and 133 in the Baerveldt group at 16 clinical centers worldwide.
Period: Overall Study
Arm/Group | Ahmed Implant,1 | Baerveldt Implant
Started | 143 | 133
Completed | 87 | 87
Not Completed | 56 | 46

BASELINE CHARACTERISTICS:
Population: One eye of each patient will be randomized to receive either an Ahmed or a Baerveldt glaucoma drainage implant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ahmed Implant,1 | Baerveldt Implant | Total
Number analyzed (Participants) | 143 | 133 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (12.8) | 62.2 (14.2) | 63.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 63 | 133
  Male | 73 | 70 | 143

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: intraocular pressure mmHg at 5 years
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Ahmed Implant,1 | Baerveldt Implant
Number analyzed (Participants) | 87 | 87
mm Hg | 14.7 (4.4) | 12.7 (4.5)

2. Primary Outcome: Failure Rate
Description: 5-year failure rate measured by Kaplan-Meier, defined as IOP>21 mm Hg or less than a 20% reduction below baseline on 2 consecutive study visits after 3 months, reoperation for glaucoma, loss of light perception, or removal of implant
Time Frame: 5 years
Population: Kaplan-Meier survival analysis
Measure: Number; unit: percent fail
Arm/Group | Ahmed Implant,1 | Baerveldt Implant
Number analyzed (Participants) | 143 | 133
percent fail | 80 | 53

3. Secondary Outcome: Visual Acuity
Description: Snellen chart converted to logMAR (smaller logMAR values indicate better visual acuity logMar of 0 is Snellen 20/20; logMAR of 20/200 is 1.0)
Time Frame: 5 years
Population: The failure rate is based on Kaplan Meier analysis of all patients enrolled (n=276).
  The five-year intraocular pressure and visual acuity outcomes are based on those patients who received a five-year visit (n=174 for IOP; n=173 for visual acuity, 1 patient had missing data)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Ahmed Implant,1 | Baerveldt Implant
Number analyzed (Participants) | 86 | 87
logMAR | 1.42 (1.15) | 1.43 (1.40)

ADVERSE EVENTS:
Time Frame: 5 year
Arm/Group | Ahmed Implant,1 | Baerveldt Implant
Serious Adverse Events (participants affected / at risk) | 9/143 | 16/133
Other Adverse Events (participants affected / at risk) | 30/143 | 29/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ahmed Implant,1 (N=143) | Baerveldt Implant (N=133)
loss of light perception (Eye disorders) | 9 | 16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ahmed Implant,1 (N=143) | Baerveldt Implant (N=133)
diplopia (Eye disorders) | 16 | 14
corneal edema (Eye disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No